CLINICAL TRIAL: NCT01696968
Title: Prostate, Lung, Colorectal, and Ovarian (PLCO) Cancer Screening Trial
Brief Title: Screening for Lung Cancer in Older Patients (PLCO Screening Trial)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: NCI-2012-01756; NCI-2012-01756 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000078532; NCI-P93-0050; PLCO-1; PLCO-Lung (Other: National Cancer Institute)
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — X-Rays; Phantoms, Imaging

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Control (No Intervention): Participants receive standard medical care. Participants complete a DHQ at baseline.
- Lung Screening (Active Comparator): Participants undergo a chest x-ray (one postero-anterior view) at baseline and annually for 2 years. Participants classified as "smokers" undergo an additional chest x-ray at year 3. Participants complete a BQF/M at baseline. Participants complete a DQX at baseline and DHQ at year 3. An ADU (previously referred to as the PSH questionnaire) is mailed to each participant annually for 13 years to identify all prevalent and incident lung cancers as all deaths that occur among both screened and control subjects during the trial.
  Interventions: Other: Screening Questionnaire Administration; Procedure: X-Ray Imaging

INTERVENTIONS:
Other: Screening Questionnaire Administration — Undergo questionnaire assessments
  Arms: Lung Screening
Procedure: X-Ray Imaging — Undergo a chest x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray
  Arms: Lung Screening

SUMMARY:
This clinical trial studies whether screening methods used to diagnose cancer of the prostate, lung, colon, rectum, or ovaries can reduce deaths from these cancers. Screening tests may help doctors find cancer cells early and plan better treatment for lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether screening with chest x-ray can reduce mortality from lung cancer in women and men aged 55-74 at entry.

SECONDARY OBJECTIVES:

I. To assess screening variables, other than mortality, for each of the interventions including sensitivity, specificity, and positive predictive value.

II. To assess the incidence, stage, and survival of cancer cases. III. To investigate the mortality predictive value of biologic and/or prognostic characterizations of tumor tissue as intermediate endpoints.

IV. To conduct biomolecular and genetic research into factors associated with cancer carcinogenesis and promotion, as well as the early detection of these factors.

OUTLINE: Participants in the overall PLCO study are stratified by screening center, gender, and age (55-59 vs 60-64 vs 65-69 vs 70-74). Participants are randomized to 1 of 2 arms (control vs screening).

ARM I (Control): Participants receive standard medical care. Participants complete a Diet History Questionnaire (DHQ) at baseline.

ARM II (Lung Screening): Participants undergo a chest x-ray (one postero-anterior view) at baseline and annually for 2 years. Participants classified as "smokers" undergo an additional chest x-ray at year 3. A scheduling and tracking procedure is implemented to ensure regular attendance at repeat screens for participants screened negative or for those who are designated suspicious or positive at screening but for whom subsequent diagnostic procedures do not reveal lung cancer (follow-up diagnostic procedures are through their own medical care environment). Participants diagnosed with lung cancer via a screening test are referred for treatment in accordance with current accepted practice for appropriate stage of disease, patient age, and medical condition; a procedure is provided for contact with qualified medical personnel to insure appropriate therapy.

Participants complete a Baseline Questionnaire (BQF/M) to assess smoking status. Participants complete a Dietary Questionnaire (DQX) at baseline and DHQ at year 3. An Annual Study Update (ADU) (previously referred to as the Periodic Survey of Health [PSH] questionnaire) is mailed to each participant annually for 13 years to identify all prevalent and incident lung cancers as all deaths that occur among both screened and control subjects during the trial.

After completion of screening, participants are followed up for at least 13 years.

ELIGIBILITY:
Exclusion Criteria:

* Men and women who at the time of randomization are less than 55 or greater than or equal to 75 years of age
* Individuals undergoing treatment for cancer at this time, excluding basal-cell and squamous-cell skin cancer
* Individuals with known prior cancer of the colon, rectum, lung, prostate (men only) or ovary (women only)

  * This includes primary or metastatic PLCO cancers
* Individuals with previous surgical removal of the entire colon, one lung, or the entire prostate (men only)

  * Until October 1996, women with previous surgical removal of both ovaries were excluded from the trial. In order to increase the enrollment of women into the trial, beginning in October 1996, these women were no longer excluded for this reason.
* Individuals who are participating in another cancer screening or cancer primary prevention trial
* Males who have taken Proscar/Propecia/finasteride in the past 6 months

  * NOTE: Individuals who are already enrolled in the trial when their physician prescribes finasteride are not prevented from taking this medication. As a result, these participants will continue to be screened and followed just as those participants who are not on finasteride.
  * NOTE: Men who are taking Tamoxifen are not excluded from any part of the PLCO Screening Trial.
  * Prior to April 1, 1999 women were excluded from the trial if they were currently taking or had taken Tamoxifen or Evista\Raloxifene in the past 6 months. As of April 1999 based on a decision from the PLCO Ovary Subcommittee, women who have or are currently taking Tamoxifen or Evista\Raloxifene are not excluded from participation.
* Individuals who are unwilling or unable to sign the informed consent form
* Males who have had more than one PSA blood test in the past three years
* Individuals who have had a colonoscopy, sigmoidoscopy, or barium enema in the past three years

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154901 (Actual)
Dates: Start 1993-11-16 (Actual); Primary Completion 2012-05-21 (Actual); Study Completion 2026-03-25 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christine D Berg, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Malcomson FC, Shams-White MM, Reedy J, Huang WY, Moore SC, Loftfield E. Adherence to the 2018 World Cancer Research Fund/American Institute for Cancer Research Cancer Prevention Recommendations and risk of lifestyle-related cancers in the prostate, lung, colorectal, and ovarian cancer screening trial. BJC Rep. 2025 Nov 19;3(1):81. doi: 10.1038/s44276-025-00195-6. PMID 41261199
- [Derived] Fan Z, Zhang Y, Yao Q, Liu X, Duan H, Liu Y, Sheng C, Lyu Z, Yang L, Song F, Huang Y, Song F. Effects of joint screening for prostate, lung, colorectal, and ovarian cancer - results from a controlled trial. Front Oncol. 2024 Apr 29;14:1322044. doi: 10.3389/fonc.2024.1322044. eCollection 2024. PMID 38741776
- [Derived] You D, Wang D, Wu Y, Chen X, Shao F, Wei Y, Zhang R, Lange T, Ma H, Xu H, Hu Z, Christiani DC, Shen H, Chen F, Zhao Y. Associations of genetic risk, BMI trajectories, and the risk of non-small cell lung cancer: a population-based cohort study. BMC Med. 2022 Jun 6;20(1):203. doi: 10.1186/s12916-022-02400-6. PMID 35658861
- [Derived] Jiang Y, Xie Q, Chen R. Breast Cancer Incidence and Mortality in Relation to Hormone Replacement Therapy Use Among Postmenopausal Women: Results From a Prospective Cohort Study. Clin Breast Cancer. 2022 Feb;22(2):e206-e213. doi: 10.1016/j.clbc.2021.06.010. Epub 2021 Jun 26. PMID 34548240
- [Derived] Wang K, Wu Q, Li Z, Reger MK, Xiong Y, Zhong G, Li Q, Zhang X, Li H, Foukakis T, Xiang T, Zhang J, Ren G. Vitamin K intake and breast cancer incidence and death: results from a prospective cohort study. Clin Nutr. 2021 May;40(5):3370-3378. doi: 10.1016/j.clnu.2020.11.009. Epub 2020 Nov 16. PMID 33277073

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between November 1993 and July 2001 at 10 study centers. Recruitment was done for all four outcomes of the study (prostate, lung, colorectal and ovarian).
Pre-assignment Details: Participants signed a study informed consent prior to being randomized to a study arm.
Groups:
- Control: Participants receive standard medical care.
- Lung Screening: Participants undergo a chest x-ray (postero-anterior view chest radiograph) at baseline and annually for 2 years. Participants classified as "smokers" undergo an additional chest x-ray at year 3.
Period: Overall Study
Arm/Group | Control | Lung Screening
Started | 77456 | 77445
Completed | 76255 | 70633
Not Completed | 1201 | 6812
Not completed — Cancer Before Rand. (Lung Screening) | 0 | 8
Not completed — Died Before Randomization | 3 | 8
Not completed — Died Before ASU (Control) | 278 | 0
Not completed — Refused ASU (Control) | 920 | 0
Not completed — Refused Screen (Lung Screening) | 0 | 6796

BASELINE CHARACTERISTICS:
Groups:
- Lung Screening: Participants undergo a chest x-ray (one postero-anterior view) at baseline and annually for 2 years. Participants classified as "smokers" undergo an additional chest x-ray at year 3.
- Total: Total of all reporting groups
Arm/Group | Control | Lung Screening | Total
Number analyzed (Participants) | 77456 | 77445 | 154901
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49612 | 49634 | 99246
  >=65 years | 27844 | 27811 | 55655
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (5.4) | 62.6 (5.4) | 62.6 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39111 | 39105 | 78216
  Male | 38345 | 38340 | 76685
Region of Enrollment [Number; unit: participants]
  United States | 77456 | 77445 | 154901

OUTCOME MEASURES:

1. Primary Outcome: Lung Cancer Deaths
Description: Lung cancer deaths confirmed in participants by a death review committee if available, otherwise by death certificate.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 11.9 years.
Population: All participants were analyzed. An intention-to-treat analysis was performed.
Measure: Number; unit: Participants
Arm/Group | Control | Lung Screening
Number analyzed (Participants) | 77456 | 77445
Participants | 1230 | 1213
Statistical Analysis 1: Comparison: Control vs Lung Screening; Test type: Superiority or Other; Poisson regression; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.91 to 1.07]

2. Secondary Outcome: Deaths From All Causes
Description: Deaths from all causes were compared between the lung screening arm and the usual care arm.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 11.9 years.
Population: All participants were analyzed. An intention-to-treat analysis was performed.
Measure: Number; unit: Participants
Arm/Group | Control | Lung Screening
Number analyzed (Participants) | 77456 | 77445
Participants | 11061 | 10827

3. Secondary Outcome: Death Rates From All Causes
Description: Deaths from all causes were compared between the lung screening arm and the usual care arm. Rate is the number of deaths divided by person years of follow-up in the study.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 11.9 years.
Population: All participants were analyzed. An intention-to-treat analysis was performed.
Measure: Number; unit: Deaths per 10,000 PY
Arm/Group | Control | Lung Screening
Number analyzed (Participants) | 77456 | 77445
Deaths per 10,000 PY | 128.1 | 125.3
Statistical Analysis 1: Comparison: Control vs Lung Screening; Test type: Superiority or Other; Poisson regression; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.95 to 1.00]

4. Secondary Outcome: Lung Cancer Incidence
Description: Lung cancer diagnoses confirmed by medical record abstraction.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 11.9 years.
Population: All participants were analyzed. An intention-to-treat analysis was performed.
Measure: Number; unit: Participants
Arm/Group | Control | Lung Screening
Number analyzed (Participants) | 77456 | 77445
Participants | 1620 | 1696

5. Secondary Outcome: Lung Cancer Incidence Rates
Description: Lung cancer diagnoses confirmed by medical record abstraction. Incidence rate (cumulative) defined as lung cancer diagnoses divided by person years at risk for lung cancer.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 11.9 years.
Population: All participants were analyzed. An intention-to-treat analysis was performed.
Measure: Number; unit: Diagnoses per 10,000 PY
Arm/Group | Control | Lung Screening
Number analyzed (Participants) | 77456 | 77445
Diagnoses per 10,000 PY | 19.2 | 20.1
Statistical Analysis 1: Comparison: Control vs Lung Screening; Test type: Superiority or Other; Poisson regression; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.98 to 1.12]

6. Secondary Outcome: Complications of Diagnostic Evaluation Following a Positive Screening Test
Description: Number of positive screens with complications.
Time Frame: One year from screening examination
Population: The units analyzed were positive screening exams with documented diagnostic follow-up. If a participant received 3 positive screens with documented follow-up after each one, he would be counted 3 times in the number of units analyzed.
Measure: Number; unit: Positive screens w/ complications
Units Other Than Participants: Positive Screens with Follow-up
Arm/Group | Lung Screening
Number analyzed (Participants) | 12889
Number analyzed (Positive Screens with Follow-up) | 17475
Positive screens w/ complications
  When DE Led to Lung Cancer Diagnosis | 173
  When DE Did Not Lead to Lung Cancer Diagnosis | 72

7. Secondary Outcome: T0 (Baseline) CXR Screening Results
Description: Postero-anterior view chest radiograph (CXR) result
Time Frame: T0 (at study entry)
Population: All participants in the Lung Screening arm who had a CXR screen at T0 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Lung Screening
Number analyzed (Participants) | 67037
Participants
  Negative | 61009
  Positive | 5965
  Inadequate screen | 63

8. Secondary Outcome: T1 CXR Screening Results
Description: Postero-anterior view chest radiograph (CXR) result
Time Frame: T1 (one year after entry)
Population: All participants in the Lung Screening arm who had a CXR screen at T1 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Lung Screening
Number analyzed (Participants) | 64706
Participants
  Negative | 60015
  Positive | 4614
  Inadequate screen | 77

9. Primary Outcome: Lung Cancer Death Rates
Description: Lung cancer deaths confirmed in participants by a death review committee if available, otherwise by death certificate. Rate is the number of deaths divided by person years of follow-up in the study.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 11.9 years.
Measure: Number; unit: Deaths per 10,000 PY
Arm/Group | Control | Lung Screening
Number analyzed (Participants) | 77456 | 77445
Deaths per 10,000 PY | 14.2 | 14.0
Statistical Analysis 1: Comparison: Control vs Lung Screening; Test type: Superiority or Other; Poisson regression; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.91 to 1.07]

10. Secondary Outcome: T2 CXR Screening Results
Description: Postero-anterior view chest radiograph (CXR) result
Time Frame: T2 (two years after entry)
Population: All participants in the Lung Screening arm who had a CXR screen at T2 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Lung Screening
Number analyzed (Participants) | 63305
Participants
  Negative | 59080
  Positive | 4157
  Inadequate screen | 68

11. Secondary Outcome: T3 CXR Screening Results
Description: Postero-anterior view chest radiograph (CXR) result
Time Frame: T3 (three years after entry)
Population: All participants in the Lung Screening arm who had a CXR screen at T3 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Lung Screening
Number analyzed (Participants) | 41403
Participants
  Negative | 38450
  Positive | 2908
  Inadequate screen | 45

ADVERSE EVENTS:
Time Frame: During each annual screening visit.
Description: These events are solely those prompted by the screening examination.
Arm/Group | Lung Screening
Serious Adverse Events (participants affected / at risk) | 0/77445
Other Adverse Events (participants affected / at risk) | 0/77445

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less